CLINICAL TRIAL: NCT03047330
Title: Menopausal Sleep Fragmentation: Impact on Body Fat Gain Biomarkers in Women
Brief Title: Menopausal Sleep Fragmentation and Body Fat Gain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hadine Joffe, MD MSc, Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P002821; 1R01AG053838 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-02-08 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Menopause
Keywords: menopause; sleep fragmentation; leuprolide; adipokine; weight gain; leptin
MeSH Terms: conditions — Sleep Deprivation; Weight Gain | interventions — Leuprolide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Participants completed 2 nights of unfragmented sleep followed by 3 nights of experimentally-fragmented sleep during high estradiol (E2) phase of their menstrual cycle (Sleep Block 1). A subset of participants repeated these procedures in an experimentally-induced low-E2 state (Sleep Block 2).
  Interventions: Drug: Estradiol withdrawal; Other: Fragmented sleep

INTERVENTIONS:
Drug: Estradiol withdrawal — one injection of open-label intramuscular dose of leuprolide (3.75-mg depot), a gonadotropin-releasing hormone agonist that rapidly suppresses estradiol and temporarily achieves ovarian suppression.
  Other Names: Leuprolide Acetate; Lupron
Other: Fragmented sleep — Fragmented sleep will be experimentally induced.

SUMMARY:
This study aims to investigate the impact of menopause-related sleep fragmentation on metabolic biomarkers of body fat gain. The investigators hypothesize that experimental sleep fragmentation will result in an adverse leptin response as a metabolic biomarker for body fat gain.

DETAILED DESCRIPTION:
While obesity is highly prevalent in midlife and older women, with rates increasing markedly after age 40 and body fat increasing in half of women during and after the menopause transition, factors causing these changes are not well understood. Reduced total sleep time has been shown to adversely impact biomarkers of obesity, but the effect of the highly prevalent menopause-related sleep fragmentation secondary to hot flashes on metabolism and eating behaviors in humans is not known. We will use experimental paradigms to isolate the impact of menopause-related sleep disruption, as well as that of hot flashes and estrogen withdrawal, metabolic biomarkers of body fat gain and on eating behaviors, results of which will inform strategies to prevent body fat gain and improve cardio-metabolic health outcomes in women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal women 18-45 years old
* Regular sleep schedule
* Limited alcohol and caffeine intake
* Regular monthly menstrual cycles
* No lifetime history of hot flashes
* Willingness to use approved methods of contraception during study
* Not obese
* Good general health

Exclusion Criteria:

* Contraindication, hypersensitivity or previous adverse reaction to gonadotropin releasing hormone agonists
* Pregnancy
* Breastfeeding
* Tobacco use
* Contraindicated systemic hormone medications or centrally active medications
* Shift workers or recent/expected time zone travel
* Obstructive sleep apnea
* Insomnia symptoms
* Diagnosis of osteoporosis or osteopenia
* Hypothalamic-pituitary-adrenal axis disorders
* Diabetes
* Gastric bypass, metabolic disorders, or other related conditions
* Abnormalities on screening laboratory tests
* Substantial hearing impairment
* Cardiovascular illness
* Neurological illness
* Recent psychiatric illness or substance-use disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: All participants who initiated Sleep Block 1
Period: Sleep Block 1
Arm/Group | Study Arm
Started | 41
Completed | 38
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Sleep Block 2
Arm/Group | Study Arm
Started | 27 (11 participants withdrew after completing Sleep Block 1 but before completing Sleep Block 2.)
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Study Arm: All participants who completed Sleep Block 1
Arm/Group | Baseline Study Arm
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 22
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Normalized Serum Leptin Levels
Description: 12-hr overnight fasted AM (morning) blood samples were assayed for leptin levels on study days 2-6 under both estrogenized and estradiol-withdrawal conditions [total: 10 samples]. For each individual, leptin values were normalized relative to the mean baseline leptin value. Baseline was defined as the unfragmented estrogenized condition (avg. of study days 2-3 in the estrogenized condition).
Time Frame: pre/post sleep fragmentation (3 days); pre/post estradiol withdrawal (~5 weeks)
Population: To compare between study conditions, leptin levels [12-hr overnight fasted AM samples] were averaged across 2 samples [on study days 2-3] before 2 nights of sleep fragmentation and across 3 samples [on study days 4-6] after 3 nights of sleep fragmentation. Leptin levels were averaged across 5 samples [on study days 2-6] ~1 week before leuprolide administration (pre-estradiol withdrawal) and across 5 samples [on study days 2-6] ~4 weeks after leuprolide administration (post-estradiol withdrawal)
Measure: Mean (Standard Error); unit: percentage of mean baseline leptin
Groups:
- Sleep Fragmentation - Active: Participants after 3 nights of experimentally-fragmented sleep
  Fragmented sleep: Fragmented sleep will be experimentally induced.
- Sleep Fragmentation - Control: Participants after 2 nights of unfragmented sleep
- Estradiol Withdrawal - Active: Participants after experimentally-induced hypo-estradiol
  Estradiol withdrawal: one injection of open-label intramuscular dose of leuprolide (3.75-mg depot), a gonadotropin-releasing hormone agonist that rapidly suppresses estradiol and temporarily achieves ovarian suppression.
- Estradiol Withdrawal - Control: Participants during high-estradiol phase of menstrual cycle
Arm/Group | Sleep Fragmentation - Active | Sleep Fragmentation - Control | Estradiol Withdrawal - Active | Estradiol Withdrawal - Control
Number analyzed (Participants) | 38 | 38 | 27 | 38
percentage of mean baseline leptin | 96.7 (2.5) | 94.0 (1.5) | 90.0 (3.0) | 101.0 (1.1)
Statistical Analysis 1: Comparison: Sleep Fragmentation - Active vs Sleep Fragmentation - Control; Test type: Superiority; p = 0.22, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol Withdrawal - Active vs Estradiol Withdrawal - Control; Test type: Superiority; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Normalized Satiety Scores
Description: 12-hr overnight fasted AM satiety scores were collected on study days 2-6 under both estrogenized and estradiol-withdrawal conditions [total: 10 scores]. For each individual, satiety scores were normalized relative to the mean baseline satiety score. Baseline was defined as the unfragmented estrogenized condition (avg. of study days 2-3 in the estrogenized condition).
Time Frame: pre/post sleep fragmentation (3 days); pre/post estradiol withdrawal (~5 weeks)
Population: To compare between study conditions, satiety scores [12-hr overnight fasted AM satiety scores] were averaged across 2 scores [on study days 2-3] before sleep fragmentation and across 3 scores [on study days 4-6] after 3 nights of sleep fragmentation. Satiety scores were averaged across 5 scores [on study days 2-6] ~1 week before leuprolide administration (pre-estradiol withdrawal) and across 5 scores [on study days 2-6] ~4 weeks after leuprolide administration (post-estradiol withdrawal).
Measure: Mean (Standard Error); unit: percentage of mean baseline satiety
Arm/Group | Sleep Fragmentation - Active | Sleep Fragmentation - Control | Estradiol Withdrawal - Active | Estradiol Withdrawal - Control
Number analyzed (Participants) | 38 | 38 | 27 | 38
percentage of mean baseline satiety | 99.2 (11.9) | 113.1 (11.0) | 102.6 (15.6) | 109.3 (7.8)
Statistical Analysis 1: Comparison: Sleep Fragmentation - Active vs Sleep Fragmentation - Control; Test type: Superiority; p = 0.048, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol Withdrawal - Active vs Estradiol Withdrawal - Control; Test type: Superiority; p = 0.58, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 4 months
Description: Since participants received interventions simultaneously, it was not possible to attribute adverse events to any one intervention. Therefore, adverse events are presented for the larger group of all participants who initiated study procedures.
Groups:
- All Participants: All participants who initiated study procedures
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 32/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=41)
Fatigue (General disorders) | 3 (3)
Gastrointestional disturbance (Gastrointestinal disorders) | 7 (7)
Headache (Nervous system disorders) | 15 (15)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4)
Skin discomfort/irritation (Skin and subcutaneous tissue disorders) | 18 (18)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 5 (5)
Amenorrhea (Reproductive system and breast disorders) | 3 (3)
Menstrual (Reproductive system and breast disorders) | 4 (4)
Vasomotor symptoms (Reproductive system and breast disorders) | 25 (25)
IV discomfort/irritation (Injury, poisoning and procedural complications) | 13 (13)
Dizziness (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03047330/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03047330/SAP_001.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03047330/ICF_003.pdf